CLINICAL TRIAL: NCT01721889
Title: Radiostereometric Analysis of Spine Arthrodesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OAD Orthopaedics (Other)
Collaborators: Halifax Biomedical Inc. (Industry); Central DuPage Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RSA100
Record Dates: First submitted 2012-10-31; First posted 2012-11-06 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Radiostereometric analysis - Intact fusion: Clinically fused per classical radiographic assessment (≤ 2 degrees angular motion and evidence of bone bridging)
  Interventions: Radiation: Radiostereometric Analysis
- Radiostereometric analysis - Symptomatic pseudoarthrosis: Definitive clinical evidence of pseudarthrosis (not fused, ˃ 2 degrees angular motion or absence of bone bridge) and scheduled for surgical exploration
  Interventions: Radiation: Radiostereometric Analysis
- Radiostereometric analysis - Asymptomatic pseudoarthrosis: Definitive clinical evidence of pseudarthrosis without scheduled surgical exploration.
  Interventions: Radiation: Radiostereometric Analysis

INTERVENTIONS:
Radiation: Radiostereometric Analysis — The radiostereometric (RSA) patient exam (flexion and extension RSA images) presents additional radiation exposure to the patient above standard of care (additional radiographs). Assuming 120kV, using three protocols (two loaded and one unloaded) per RSA exam results in a typical effective dose of approximately 2.04mSv per exam(single lumbar spine RSA at 120kV yields 0.68mSv,). HBI recommends using 140kV for lumbar spine RSA and has conducted simulations to estimate the effective dose using higher kV settings. 140kV reduces the effective dose from 0.68mSv per spine RSA to 0.2mSV, resulting in a total effective dose per RSA exam of 0.6mSv. In comparison, the estimated effective dose for a single standard lumbar spine x-ray is 1.2mSv. This additional radiation exposure is considered to be minimal risk in consideration of the number of planar x-rays the patient will undergo as part of standard care, as well as average background radiation received by humans per year (3.1mSv).

SUMMARY:
The primary objective of this pilot study is to determine the precision of post-operative radiostereometric measurements for the assessment of lumbar spinal fusion. This study will also determine the potential for RSA as a more precise and accurate means for assessment of lumbar spinal fusion and diagnosis of pseudarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic degenerative disc disease of the lumbar spine indication surgical intervention
* Scheduled to undergo lumbar fusion surgery
* Patients between the ages of 18 and 75
* Ability to give informed consent

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 75 that are diagnosed with lumbar DDD (L1-L5, and also L5-S1) and scheduled for one or multi level spinal fusion surgery will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Intervertebral motion post-op lumbar fusion | 2 years
  The purpose of this radiostereometric analysis (RSA) evaluation is to measure relative intervertebral motion in lumbar spinal fusions. Two RSA loading provocation protocols will be employed in this study; sitting and supine extension. Both loading protocols will be compard to a standard supine position which is used as an unloaded baseline protocol. Induced intervetebral motion sets will be calculated between the two loaded states, sitting and supine extension, and the unloaded state. The RSA micromotion results will be calculated and reported as translations and rotations about the three anatomic axes, maximum total point motion (MTPM) will be calculated as well.

CONTACTS AND LOCATIONS:
Overall Officials: John Andreshak, MD, Principal Investigator — OAD Orthopaedics
Locations (1):
- OAD Orthopaedics, Warrenville, Illinois, United States